CLINICAL TRIAL: NCT05007093
Title: An Exploratory Study on Efficacy of Anlotinib Hydrochloride in the Treatment of Locally Advanced or Metastatic Differentiated Thyroid Cancer
Brief Title: Study on the Treatment of Differentiated Thyroid Carcinoma with Anlotinib
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yansong Lin (Other)
Responsible Party: Sponsor-Investigator, Yansong Lin, Prof. M.D., Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EXPLORE-001
Record Dates: First submitted 2021-08-09; First posted 2021-08-16 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: DTC - Differentiated Thyroid Cancer
Keywords: Anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anlotinib hydrochloride (Experimental): 12 mg, 2 weeks on/ 1 week off, 21 days per cycle; treatment interruption or reduction (to 10 mg or 8 mg) was allowed
  Interventions: Drug: Anlotinib hydrochloride

INTERVENTIONS:
Drug: Anlotinib hydrochloride — If intolerance occurs, the dose can be downregulated

SUMMARY:
The purpose of this study is to evaluate the efficacy of anlotinib in patients with locally advanced or metastatic differentiated thyroid cancer resistant to iodine therapy.

ELIGIBILITY:
Inclusion Criteria:

* locally advanced or metastatic RAIR-DTC (papillary, follicular [including Hürthle cell], and poorly differentiated) progressed within 18 months after the last treatment according to the Response Evaluation Criteria in Solid Tumors, version 1.1
* Patients with RAIR-DTC should meet at least 1 of the following conditions: (a) the tumor invaded vital organs, cannot be completely removed nor suitable for further iodine treatment, or (b) lesions do not demonstrate iodine uptake on any radioactive iodine scan, or (c) received cumulative RAI activity ≥22.3 GBq (≥600 mCi), or (d) tumors retained iodine uptake but demonstrated radiological examination confirmed disease progression within 18 months after RAI treatment.
* at least one measurable lesion on computed tomography (CT) or magnetic resonance imaging (MRI) according to RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2
* life expectancy of at least 6 months
* adequate main organ function ((a) Hemoglobin (HBG) ≥ 90g/L, (b) neutrophil count (ANC) ≥ 1.5×109/L, (c) platelet count (PLT) ≥ 80×109/L, (d) total bilirubin < 1.5×ULN (upper limit of normal), (e) alanine aminotransferase (ALT) and aspartate aminotransferase AST ≤ 2.5×ULN, if accompanied by liver metastases, then ALT and AST ≤ 5 × ULN; (f) serum creatinine (Cr) ≤ 1.5 × ULN or creatinine clearance rate (CCr) ≥ 60 ml/min; (g) left ventricular ejection fraction ≥ 50% of the normal level
* Negative pregnancy test (serum or urine) within 7 days prior to enrollment for women of childbearing potential (subjects should use appropriate contraception until 6 months after the last dose)

Exclusion Criteria:

* Patients who have received external radiotherapy or iodine-131 therapy in recent 3 months, or plan to receive other systemic anti-tumor therapy or anti-tumor therapy with traditional Chinese medicine during the study period.
* Patients with other malignant tumors within 5 years or currently. Except primary cervical cancer, non-melanoma skin cancer and superficial bladder tumor.
* The toxicity of CTCAE (4.0) above grade 1 was not alleviated, excluding patients with neurotoxicity (≤ grade 2) and alopecia caused by oxaliplatin.
* With factors affecting oral administration (such as swallow, chronic diarrhea, etc.).
* Patients with pleural effusion or ascites causing respiratory syndrome (CTCAE2 level above).
* Patients who underwent major surgery, open biopsy or significant traumatic injury within 4 weeks.
* Regardless of the severity, patients with any physical signs or history of bleeding, patients with bleeding or bleeding events greater than or equal to CTCAE 3 within four weeks prior to the first administration, or patients with unhealed wounds, fractures, ulcers.
* Patients with arterial or venous thromboembolic events occurred within 6 months, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The changes in glucose metabolism | up to 24 months
  Evaluated by maximum standard uptake value (SUVmax)

SECONDARY OUTCOMES:
Time to response (TTR) | up to 24 months
PFS | up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun D, Zhang X, Jin X, Shi C, Sun Y, Zhang Y, Liang J, Lin Y. BRAFV600E mutation is associated with better prognoses in radioactive iodine refractory thyroid cancer patients treated with multi-kinase inhibitors: a retrospective analysis of registered clinical trials. Thyroid Res. 2025 Feb 10;18(1):5. doi: 10.1186/s13044-025-00223-0. PMID 39924483